CLINICAL TRIAL: NCT01224288
Title: Dynamic Contrast Enhancement Computed Tomography for Evaluating Tumor Perfusion in Patients With Metastatic Renal Cell Carcinoma Receiving Targeted Therapies: Companion to Protocol 2010-0085
Brief Title: Dynamic Contrast Enhancement Computed Tomography for Evaluating Tumor Perfusion in Patients With Metastatic Renal Cell Carcinoma Receiving Targeted Therapies: Renal Cell Carcinoma (RCC) Scramble
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-0845; NCI-2011-03288 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Renal Cell Carcinoma
Keywords: RCC; Kidney cancer; Metastatic renal cell carcinoma; mRCC; Dynamic contrast enhanced CT; DCE-CT; Tumor perfusion
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DCE-CT Scans (Experimental): DCE-CT = Dynamic contrast enhanced CT - DCE-CT scans 4 weeks prior to and 8 weeks after starting treatment on study 2010-0085.
  Interventions: Procedure: Perfusion CT scan

INTERVENTIONS:
Procedure: Perfusion CT scan — DCE-CT scans 4 weeks prior to and 8 weeks after starting treatment on study 2010-0085.

SUMMARY:
This is a companion protocol to MD Anderson Cancer Center study 2010-0085 (Sequential Therapy in Advanced Renal Cell Carcinoma Therapy: The "START" Trial).

The goal of this clinical research study is to learn if dynamic contrast enhanced computed tomography (DCE-CT) scans can help researchers learn if the study drug received as part of study 2010-0085 (either everolimus, bevacizumab, or pazopanib) is working.

DETAILED DESCRIPTION:
To perform a DCE-CT scan, a small amount of a special dye (called "CT contrast medium") is injected by vein into the body. Several CT images are then taken over a few minutes to learn how much dye spreads outside of the tumor. This can show how much blood flows to and from the tumor. By performing DCE-CT scans after several weeks on treatment, researchers may learn if changes in blood flow may be a sign that the treatment is working.

Study Procedures:

If you are found to be eligible to take part in this study, you will have a DCE-CT scan to check the status of the disease at the following times:

* Within about 4 weeks before you begin treatment on study 2010-0085.
* Eight (8) weeks after starting treatment on study 2010-0085.

Before each of the DCE-CT scans are performed, blood (about 1 tablespoon) will be drawn to check your kidney function.

If your doctor thinks it is needed, you will also have a standard-of-care CT scan at these timepoints to check the status of the disease.

Length of Study:

Your participation in this study will be over after the scan(s) 8 weeks after starting treatment on study 2010-0085. You will be taken off of this study if you leave the 2010-0085 study early.

This is an investigational study. The DCE-CT scan is commercially available. Using DCE-CT scans to check the status of kidney cancer is investigational.

Up to 120 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be enrolled or being considered for enrollment on protocol 2010-0085.
2. Patients must have metastatic renal cell carcinoma (RCC).
3. Age >/= 18 years.
4. Subjects must have adequate renal function as defined by serum creatinine < 1.5x upper limit of normal.

Exclusion Criteria:

1. Radiotherapy: Subjects may not have received prior radiotherapy to the index lesion within 4 weeks
2. Female subjects who are pregnant or lactating.
3. Female subjects of childbearing potential (unless they have a negative serum or urine pregnancy test within 3 days prior to start of study treatment).
4. Allergy to CT contrast media requiring the administration of steroid prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-01-05 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Tumor Blood Flow (BF) Reduction | From 4 weeks prior to first dose to 8 weeks post treatment
  Changes in perfusion parameters assessed at first re-staging (approximately 8 weeks) and shortly after initiating therapy (2 - 7 days), for three different therapies using organ-directed DCE-CT tumor assessments. Tumor BF of index lesions computed using commercially available software (GE CT perfusion) using the same index lesion assessed on follow-up scans.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 3 years
  PFS is calculated from the start of the study until disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Chaan Ng, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org